CLINICAL TRIAL: NCT02399683
Title: Mucosal and Systemic Immune Modulation From Trichuris Trichiura in a Self-infected Individual
Brief Title: Immune Modulation From Trichuris Trichiura
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Principal Investigator, Christian Hvas, MD, Ph.D., University of Aarhus
Other Study IDs: Trichuris trichiura
Record Dates: First submitted 2015-03-12; First posted 2015-03-26 (Estimated); Last update posted 2016-11-21 (Estimated); Status verified 2016-11

CONDITIONS: Crohn Disease; Colitis, Ulcerative; Intestinal Helminthiasis
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative; Intestinal helminthiasis

STUDY DESIGN:
Observational Model: Case-Only
Biospecimen Retention: Samples With DNA — Blood cell and intestinal biopsies
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Trichuris trichiura eggs: One healthy volunteer
  Interventions: Biological: Trichuris trichiura eggs

INTERVENTIONS:
Biological: Trichuris trichiura eggs — Live eggs from human whipworm, Trichuris trichiura

SUMMARY:
Mucosal immunology during helminth infection

DETAILED DESCRIPTION:
The present study investigates the effects of Trichuris trichiura on human mucosal and systemic immunity in a single self-infected individual.

ELIGIBILITY:
Inclusion Criteria:

* The included volunteer is a researcher within parasitology with main focus on Trichuris trichiura and Trichiura suis. He planned to infect himself and contacted our department with the purpose of being monitored during this infection for safety (medical supervision) and research reasons. The only clinical criterion for his inclusion in the study was that he was healthy.

Exclusion Criteria:

* N/A

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A single healthy volunteer
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2012-02; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Faecal egg excretion | 30 weeks
  Weekly monitoring of fecal egg counts by microscopy

SECONDARY OUTCOMES:
Mucosal T cell associated cytokines | Week 15
  Biopsy sampling during established infection
Systemic immune parameters (eosinophilia, Subtypes of circulating T cells) | 30 weeks
  Weekly monitoring
Adverse events | 30 weeks
  The included individual was monitored clinically every week for the development of diarrhea and weight loss, and by blood samples for anemia and inflammatory parameters every other week.

CONTACTS AND LOCATIONS:
Overall Officials: Jens F Dahlerup, MD, Principal Investigator — Aarhus University Hospital